CLINICAL TRIAL: NCT04053738
Title: An Intelligent Bed To Monitor And Reduce Snoring
Brief Title: The Anti-snoring Bed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ASB
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not informed prior to going to bed whether the night would be an intervention night or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): Participants slept in the anti-snoring bed in the laboratory, but the bed did not provide any intervention
- Anti-snoring Intervention (Experimental): Participants slept in the anti-snoring bed in the laboratory, and the bed moved the trunk of the participant
  Interventions: Device: Anti-snoring bed

INTERVENTIONS:
Device: Anti-snoring bed — The mattress shape is adjusted using a custom made intelligent anti-snoring bed, which is able to detect snoring sound and change the position of the user whenever snoring occurs.
  Arms: Anti-snoring Intervention

SUMMARY:
Habitual snoring is a widespread complication. Most snorers snore predominately when sleeping in supine position. Therefore, therapeutic interventions force snorers to avoid supine position. Devices that restrict the sleeping position or raise alarms when the user obtains the supine position cause discomfort or disrupt sleep resulting in low compliance. Therefore, anti-snoring mechanisms, which lift the trunk of the user without disturbing sleep, have been proposed.

We set out to investigate whether individual interventions provided by beds with lifting mechanisms are able to stop snoring within three minutes (success rate) and whether the bed reduces the snoring index (number of total snores divided by total time in bed). In addition, we investigat whether the trunk elevation provided by the bed is interfering with the subjective sleep quality assessed using the Groningen Sleep Quality Score.

Subjects are observed for four nights (adaptation, baseline, and two intervention nights). During intervention nights, the bed lifts the trunk of the user in closed-loop manner. Subjects are divided in three groups (non-snorers, snorer group one, and snorer group two). Non-snorers are lifted by the bed at random time points during the night. In snorer group one, a stepwise increase of the bed inclination is compared with going directly to a randomly selected angle. In snorer group two, the influence of a small inclination angle (10°) and a big inclination angle (20°) is compared..

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* Pregnancy
* Previously diagnosed sleep-related breathing disorders
* Chronic lower back pain
* Heart insufficiency that might impede sleeping in supine position
* Inability to follow the procedures of the study, e.g. due to language problems

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Effect on snoring | whole night - 4 nights
  Number of episodes of snoring that are terminated by intervention.
  Snoring activity was monitored using a portable home-monitoring device (Apnea Link plus, purchased from ResMed, Switzerland). This device records oxygen saturation, nasal airflow, and breathing effort. The device comes with a software package that automatically scores the data according to the sleep scoring rules of the American Academy of Sleep Medicine (AASM). Since audio based detection has been reported to be the most reliable way of snoring detection , we also used a sound level meter (XL2 Audio and acoustic Analyzer, purchased from NTi Audio, Lichtenstein) for manual visual-audio scoring of snoring sound. The sound level meter was placed approximately in the position where you would usually expect the head of the bed partner. Manual visual-audio scoring of the data collected with the noise level meter was performed using the XL2 data explorer.

SECONDARY OUTCOMES:
Self-Reported Sleep Quality | upon awakening - 4 nights
  Subjective Sleep Quality was assessed using the standardized Groningen Sleep Quality Scale (GSQS). This questionnaire consists of 15 questions, which are to be answered with yes or no. The maximum possible score of 14 indicates a poor sleep the preceding night. Within the study, we used the original English version of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof. Dr. Dr.-Ing., Principal Investigator — University of Zurich
Locations (1):
- Sensory-Motor Systems Lab, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No